CLINICAL TRIAL: NCT04034680
Title: The TIME -Targeted Interdisciplinary Model for Evaluation and Treatment of Neuropsychiatric Symptoms - for Continuity of Care in Home Care Services
Brief Title: Targeted Interdisciplinary Model for Evaluation and Treatment of Neuropsychiatric Symptoms in Home Care Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI0303150608
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Dementia
Keywords: Behavioral symptoms; Dementia; Nevropsychiatric symptoms; Psychological symptoms; The TIME model
MeSH Terms: conditions — Dementia; Behavioral Symptoms | interventions — Time

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Who Masked: Participant
Masking Description: Participants will be masked for the study arm they are randomised to. Staff in the home care service are aware of the study arm their patients are in, while assessors that will interview home care staff by telephone are masked for study randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home care services - Intervention group (Experimental): Totally 5 municipalities (25 persons with dementia) will be included in the intervention group, and will receive training in the TIME model. This includes two hours of lectures about dementia and neuropsychiatric symptoms (NPS) and three hours of training and roleplay in using the TIME model. The staff of the home care service will receive the TIME manual and access to the TIME website with access to additional educational and information files. From each municipality, three staff members, called TIME administrators, will receive additional three hours of lectures and roleplay in TIME, and will thereafter have the responsibility for performing the intervention.
  Interventions: Other: TIME
- Home care services - Control group (Active Comparator): Totally 5 municipalities (25 persons with dementia) will be included in the Control group. The municipalities in the control group will receive the same two hours lectures about dementia and NPS as the intervention group. After the cluster RCT pilot study is ended, municipalities in the control group will receive the same three-hour lessons in the TIME as the intervention group of municipalities.
  Interventions: Other: Education-only intervention

INTERVENTIONS:
Other: TIME — The intervention of the TIME model includes two hours of lectures about dementia and NPS and three hours of training and roleplay in using TIME. The staff of the home care service will receive the TIME manual and access to the TIME website with access to additional educational materials. From each municipality, three staff members called TIME administrators, will receive additional three hours of lectures and roleplay in TIME, and will thereafter have the responsibility for performing the intervention.
  Arms: Home care services - Intervention group
Other: Education-only intervention — Staff in the home care service in municipalities in the control group will receive thesame two hours lectures about dementia and NPS as the intervention grorp. After the cluster RCT pilot study is ended, municipalities in the control group will receive the same three-hour lessons in the TIME as the intervention group of municipalities.
  Arms: Home care services - Control group

SUMMARY:
Continuity of care in home care services is necessary to facilitate the assessment and treatment of persons with dementia and cognitive failure. TIME (Targeted Interdisciplinary Model for Evaluation and Treatment of Neuropsychiatric Symptoms) is a multi-component intervention with a biopsychosocial approach, based on the theoretical framework of cognitive behavioral therapy and person-centred care. The trial is designed to assess the effects of TIME on Neuropsychiatric symptoms for persons (NPS) with dementia in home care services.

DETAILED DESCRIPTION:
The Targeted Interdisciplinary Model for Evaluation and Treatment of Neuropsychiatric Symptoms (TIME) is a multi-component intervention with a biopsychosocial approach, based on the theoretical framework of cognitive behavioral therapy and person-centred care. TIME consists of a manual based multicomponent program which includes a rigorous assessment, treatment, and the evaluation of neuropsychiatrc symptoms (NPS).

The cluster RCT will contain two parallel groups, where randomisation is performed based on clusters. One municipality is one cluster, randomized to receive either the intervention with TIME or a brief two hours education-only intervention about dementia and NPS for the control group. Totally 10 municipalities will be included. Data will be collected at baseline before randomisation and at the end of the implementing phase. Measurements at patient level are taken at baseline prior to randomization and after 6 months. The primary outcome measure is difference in change between the intervention group and the control group from baseline to follow up at 6 months in the Cornell Scale for Depression in Dementia (CSDD).

Data collection will be performed by project nurses recruited outside the home care services. They will interview the staff or family members who knows the patient best. The assessors will be blinded to the randomization of the home care services. Interviews will be done by telephone or face-to-face, depending on what is best for the person interviewed.

After the intervention focus group interviews with staff and family members will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Dementia, defined as a score of 1 or more on the Clinical Dementia Rating Scale (CDR)
* A minimum of 15 minutes of home care services per day for the last 4 weeks
* NPS, defined as a score on the NPI-NH affective subsyndrom (NPI depression + NPI anxiety) of 12 or more
* Informed consent from the participant or family or next-of-kin

Exclusion Criteria:

* Terminal disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Affective symptoms measured by the Cornell Scale for Depression in Dementia (CSDD) | 6 months
  The change from baseline of affective symptoms as defined in the Cornell Scale for Depression in Dementia (CSDD), a scale ranging from 0-38 where a higher score indicates more severe depressive symptoms.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory - nursing home version (NPI-NH): Sub syndrome anxiety and depression | 6 months
  The change from baseline in the sub syndrome affective symptoms of the single items anxiety and depression as measured with the NPI-NH. Each single item is scored from 0-12, where a higher score indicates a more severe symptom.
NPI-NH: all separate items | 6 months
  The change from baseline of the NPI-NH, scores on all the 12 items. Each single item is scored from 0-12, where a higher score indicates a more severe symptom.
NPI-NH: caregiver distress score | 6 months
  The change from baseline in caregiver distress by the NPI-NH caregiver distress score. The caregiver distress on each NPI-NH item is scored from 0-5, where a higher score indicates more severe distress
Quality of life measured by the scale QUALID | 6 months
  The change from baseline in quality of life by whitch will be assessed by the scale QUALID: Quality of life in late-stage dementia scale, a scale consisting of 11 single items scored from 1-5 (total score 11-55) where a lower score indicates a better QoL.
Change in Relatives Stress scale Score (RSS) | 6 months
  The change in relatives stress assessed by the scale RSS: Relatives Stress scale Score, a scale ranging from 0-60 where a higher score indicates more severe distress
Transferring to nursing home | 12 months
  To measure the number of patients transferring to nursing home during follow up.
Minimal data set (MDS): patient rejection of care | 6 months
  The change in the patients rejection of care assessed by MDS: Minimal dataset (MDS)

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Bergh, PhD, Principal Investigator — The Research centre for Age-related Functional decline and Disease (AFS)
Locations (1):
- The Research centre for Age-related Functional decline and Disease (AFS) at Innlandet Hospital Trust, Ottestad, Norway